CLINICAL TRIAL: NCT02942407
Title: RENal Hemodialysis Patients ALlocated Apixaban Versus Warfarin in Atrial Fibrillation (RENAL-AF) Randomized Clinical Trial
Brief Title: Trial to Evaluate Anticoagulation Therapy in Hemodialysis Patients With Atrial Fibrillation
Acronym: RENAL-AF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Christopher Granger, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Christopher Granger, MD, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00068545
Record Dates: First submitted 2016-04-14; First posted 2016-10-24 (Estimated); Results first posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Atrial Fibrillation; End Stage Renal Disease
Keywords: Renal dialysis
MeSH Terms: conditions — Atrial Fibrillation; Kidney Failure, Chronic | interventions — apixaban; Warfarin; Vitamin B 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- apixaban (Experimental): apixaban 5 mg twice daily (apixaban 2.5 mg twice daily for selected patients)
  Interventions: Drug: apixaban
- warfarin (Experimental): warfarin daily dose adjusted to target International Normalized Ration(INR) of 2-3
  Interventions: Drug: warfarin

INTERVENTIONS:
Drug: apixaban — oral anticoagulant
  Other Names: Eliquis
  Arms: apixaban
Drug: warfarin — oral anticoagulant
  Other Names: Coumadin; Jantoven
  Arms: warfarin

SUMMARY:
This is a prospective, randomized, open-label, blinded end-point evaluation trial. The patient population consists of patients on hemodialysis who have atrial fibrillation (AF) and end-stage renal disease (ESRD) .

DETAILED DESCRIPTION:
This is a multicenter study in adult patients with AF and ESRD who are on hemodialysis and who have stroke risk factors making them candidates for oral anticoagulation. Patients will be randomized to apixaban versus warfarin, and will be treated for up to 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age at least 18 years, or the local age of consent, whichever is greater.
* Patients with AF defined as AF on ECG at enrollment or two or more reports of AF from separate monitoring events at least 2 weeks apart (report of ECG, Holter monitor, event monitor or implantable loop recorder).
* CHA2DS2-VASc score of ≥ 2.
* End-stage renal disease treated with hemodialysis for ≥ 3 months.
* Considered by the treating physician(s) to be candidate for oral anticoagulation.
* If of childbearing potential, be willing to avoid pregnancy during the study.

Exclusion Criteria:

* Not considered by the treating physician(s) to be candidates for oral anticoagulation (for example, hemoglobin < 8.5g/dL, history of intracranial hemorrhage, active bleeding, recent gastrointestinal bleed or retroperitoneal bleed, severe hepatic impairment, or anaphylactic reaction to apixaban)
* Moderate or severe mitral stenosis
* Conditions other than AF that require anticoagulation such as mechanical prosthetic valve, deep venous thrombosis, or pulmonary embolism
* Need for aspirin at a dose > 81 mg a day or need for P2Y12 antagonist therapy (for example clopidogrel, prasugrel, or ticagrelor)
* Life expectancy < 3 months
* Anticipated kidney transplant within the next 3 months
* Prisoners or others who are involuntarily incarcerated or detained
* Pregnant, breastfeeding, or considering pregnancy.
* Participation in a clinical trial of an experimental treatment within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-07-27 (Actual); Study Completion 2019-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Granger, MD, Principal Investigator — Duke University; Glenn Chertow, MD, Principal Investigator — Stanford University
Locations (58):
- United States (58):
  - Nephrology Consultants, Huntsville, Alabama
  - The Medical Research Group, Inc., Fresno, California
  - DaVita Clinical Trials, LLC, Long Beach, California
  - Southland Renal Medical Group, Long Beach, California
  - Valley Renal Medical Group Research, Northridge, California
  - Summit Nephrology Medical Group, Inc., Roseville, California
  - Satellite Healthcare, San Jose, California
  - Washington Nephrology Associates, Washington D.C., District of Columbia
  - South Florida Nephrology Group PA, Research Division, Coral Springs, Florida
  - LG. Diagnostic, Inc. & Cosmetic Center, Miami, Florida
  - Nuren Medical and Research Center, Miami, Florida
  - Medical Professional Clinical Research Center, Miami, Florida
  - Boise Kidney and Hypertension Institute, Meridian, Idaho
  - Northwestern University, Chicago, Illinois
  - NANI Research, Crystal Lake, Illinois
  - NANI Research, River Forest, Illinois
  - NANI Research, Fort Wayne, Indiana
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - Anne Arundel Medical Center, Annapolis, Maryland
  - The Johns Hopkins University, Baltimore, Maryland
  - Washington Nephrology Associates, Takoma Park, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - South Shore Nephrology, Plymouth, Massachusetts
  - Renal and Transplant Associates of New England, Springfield, Massachusetts
  - Paragon Health Neprhology Centre, Kalamazoo, Michigan
  - St. Clair Nephrology, Port Huron, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Southwest Mississippi Nephrology, PLLC, Brookhaven, Mississippi
  - Southern Clinical Research Group, LLC, Gulfport, Mississippi
  - Nephrology & Hypertension Associates, Tupelo, Mississippi
  - Polack Renal, LLC, St Louis, Missouri
  - Sierra Nevada Nephrology Consultants, Reno, Nevada
  - Renal Medicine Associates, Albuquerque, New Mexico
  - Advanced Kidney Care of Hudson Valley, Poughkeepsie, New York
  - Durham Nephrology Associates, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Eastern Nephrology Associates, PLLC., Kinston, North Carolina
  - Eastern Nephrology Associates, PLLC, New Bern, North Carolina
  - HNC Dialysis, Ltd., Columbus, Ohio
  - Northeast Clinical Research Ctr, Bethlehem, Pennsylvania
  - Penn State Health - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Columbia Nephrology Associates, Columbia, South Carolina
  - South Carolina Nephrology and Hypertension, Orangeburg, South Carolina
  - Sumter Medical Specialists, Sumter, South Carolina
  - Regional Health Clinical Research, Rapid City, South Dakota
  - Knoxville Kidney Center, Knoxville, Tennessee
  - Southwest Houston Research, Ltd., Houston, Texas
  - Lubbock Vascular Access Center, Lubbock, Texas
  - University of Utah, Salt Lake City, Utah
  - Washington Nephrology Associates, Alexandria, Virginia
  - University of Virgina Health System, Charlottesville, Virginia
  - TPMG Clinical Research, Newport News, Virginia
  - Valley Nephrology Associates, Roanoke, Virginia
  - University of Washington, Seattle, Washington
  - Nephrology and Hypertension Associates, Bluefield, West Virginia
  - West Virginia University, Morgantown, West Virginia
  - Aspirius Research Institute, Wausau, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wizemann V, Tong L, Satayathum S, Disney A, Akiba T, Fissell RB, Kerr PG, Young EW, Robinson BM. Atrial fibrillation in hemodialysis patients: clinical features and associations with anticoagulant therapy. Kidney Int. 2010 Jun;77(12):1098-106. doi: 10.1038/ki.2009.477. Epub 2010 Jan 6. PMID 20054291
- [Background] Olesen JB, Lip GY, Kamper AL, Hommel K, Kober L, Lane DA, Lindhardsen J, Gislason GH, Torp-Pedersen C. Stroke and bleeding in atrial fibrillation with chronic kidney disease. N Engl J Med. 2012 Aug 16;367(7):625-35. doi: 10.1056/NEJMoa1105594. PMID 22894575
- [Background] Nigwekar SU, Bhan I, Turchin A, Skentzos SC, Hajhosseiny R, Steele D, Nazarian RM, Wenger J, Parikh S, Karumanchi A, Thadhani R. Statin use and calcific uremic arteriolopathy: a matched case-control study. Am J Nephrol. 2013;37(4):325-32. doi: 10.1159/000348806. Epub 2013 Mar 21. PMID 23548843
- [Background] Yang F, Chou D, Schweitzer P, Hanon S. Warfarin in haemodialysis patients with atrial fibrillation: what benefit? Europace. 2010 Dec;12(12):1666-72. doi: 10.1093/europace/euq387. Epub 2010 Nov 2. PMID 21045011
- [Background] Chan KE, Lazarus JM, Thadhani R, Hakim RM. Warfarin use associates with increased risk for stroke in hemodialysis patients with atrial fibrillation. J Am Soc Nephrol. 2009 Oct;20(10):2223-33. doi: 10.1681/ASN.2009030319. Epub 2009 Aug 27. PMID 19713308
- [Background] Shah M, Avgil Tsadok M, Jackevicius CA, Essebag V, Eisenberg MJ, Rahme E, Humphries KH, Tu JV, Behlouli H, Guo H, Pilote L. Warfarin use and the risk for stroke and bleeding in patients with atrial fibrillation undergoing dialysis. Circulation. 2014 Mar 18;129(11):1196-203. doi: 10.1161/CIRCULATIONAHA.113.004777. Epub 2014 Jan 22. PMID 24452752
- [Background] Granger CB, Chertow GM. A pint of sweat will save a gallon of blood: a call for randomized trials of anticoagulation in end-stage renal disease. Circulation. 2014 Mar 18;129(11):1190-2. doi: 10.1161/CIRCULATIONAHA.113.007549. Epub 2014 Jan 22. No abstract available. PMID 24452751
- [Background] Chan KE, Edelman ER, Wenger JB, Thadhani RI, Maddux FW. Dabigatran and rivaroxaban use in atrial fibrillation patients on hemodialysis. Circulation. 2015 Mar 17;131(11):972-9. doi: 10.1161/CIRCULATIONAHA.114.014113. Epub 2015 Jan 16. PMID 25595139
- [Background] Hart RG, Pearce LA, Asinger RW, Herzog CA. Warfarin in atrial fibrillation patients with moderate chronic kidney disease. Clin J Am Soc Nephrol. 2011 Nov;6(11):2599-604. doi: 10.2215/CJN.02400311. Epub 2011 Sep 8. PMID 21903982
- [Background] Reinecke H, Brand E, Mesters R, Schabitz WR, Fisher M, Pavenstadt H, Breithardt G. Dilemmas in the management of atrial fibrillation in chronic kidney disease. J Am Soc Nephrol. 2009 Apr;20(4):705-11. doi: 10.1681/ASN.2007111207. Epub 2008 Dec 17. PMID 19092127
- [Background] Hart RG, Pearce LA, Aguilar MI. Meta-analysis: antithrombotic therapy to prevent stroke in patients who have nonvalvular atrial fibrillation. Ann Intern Med. 2007 Jun 19;146(12):857-67. doi: 10.7326/0003-4819-146-12-200706190-00007. PMID 17577005
- [Background] Winkelmayer WC, Liu J, Setoguchi S, Choudhry NK. Effectiveness and safety of warfarin initiation in older hemodialysis patients with incident atrial fibrillation. Clin J Am Soc Nephrol. 2011 Nov;6(11):2662-8. doi: 10.2215/CJN.04550511. Epub 2011 Sep 29. PMID 21959598
- [Background] Hohnloser SH, Hijazi Z, Thomas L, Alexander JH, Amerena J, Hanna M, Keltai M, Lanas F, Lopes RD, Lopez-Sendon J, Granger CB, Wallentin L. Efficacy of apixaban when compared with warfarin in relation to renal function in patients with atrial fibrillation: insights from the ARISTOTLE trial. Eur Heart J. 2012 Nov;33(22):2821-30. doi: 10.1093/eurheartj/ehs274. Epub 2012 Aug 29. PMID 22933567
- [Background] Elliott MJ, Zimmerman D, Holden RM. Warfarin anticoagulation in hemodialysis patients: a systematic review of bleeding rates. Am J Kidney Dis. 2007 Sep;50(3):433-40. doi: 10.1053/j.ajkd.2007.06.017. PMID 17720522
- [Background] Wu JR, DeWalt DA, Baker DW, Schillinger D, Ruo B, Bibbins-Domingo K, Macabasco-O'Connell A, Holmes GM, Broucksou KA, Erman B, Hawk V, Cene CW, Jones CD, Pignone M. A single-item self-report medication adherence question predicts hospitalisation and death in patients with heart failure. J Clin Nurs. 2014 Sep;23(17-18):2554-64. doi: 10.1111/jocn.12471. Epub 2013 Dec 20. PMID 24355060
- [Background] Gonzalez JS, Schneider HE, Wexler DJ, Psaros C, Delahanty LM, Cagliero E, Safren SA. Validity of medication adherence self-reports in adults with type 2 diabetes. Diabetes Care. 2013 Apr;36(4):831-7. doi: 10.2337/dc12-0410. Epub 2012 Nov 30. PMID 23204245
- [Background] Halvorsen S, Atar D, Yang H, De Caterina R, Erol C, Garcia D, Granger CB, Hanna M, Held C, Husted S, Hylek EM, Jansky P, Lopes RD, Ruzyllo W, Thomas L, Wallentin L. Efficacy and safety of apixaban compared with warfarin according to age for stroke prevention in atrial fibrillation: observations from the ARISTOTLE trial. Eur Heart J. 2014 Jul 21;35(28):1864-72. doi: 10.1093/eurheartj/ehu046. Epub 2014 Feb 20. PMID 24561548
- [Background] Fox KA, Piccini JP, Wojdyla D, Becker RC, Halperin JL, Nessel CC, Paolini JF, Hankey GJ, Mahaffey KW, Patel MR, Singer DE, Califf RM. Prevention of stroke and systemic embolism with rivaroxaban compared with warfarin in patients with non-valvular atrial fibrillation and moderate renal impairment. Eur Heart J. 2011 Oct;32(19):2387-94. doi: 10.1093/eurheartj/ehr342. Epub 2011 Aug 28. PMID 21873708
- [Background] Farrington CP, Manning G. Test statistics and sample size formulae for comparative binomial trials with null hypothesis of non-zero risk difference or non-unity relative risk. Stat Med. 1990 Dec;9(12):1447-54. doi: 10.1002/sim.4780091208. PMID 2281232
- [Background] Connolly SJ, Eikelboom J, Joyner C, Diener HC, Hart R, Golitsyn S, Flaker G, Avezum A, Hohnloser SH, Diaz R, Talajic M, Zhu J, Pais P, Budaj A, Parkhomenko A, Jansky P, Commerford P, Tan RS, Sim KH, Lewis BS, Van Mieghem W, Lip GY, Kim JH, Lanas-Zanetti F, Gonzalez-Hermosillo A, Dans AL, Munawar M, O'Donnell M, Lawrence J, Lewis G, Afzal R, Yusuf S; AVERROES Steering Committee and Investigators. Apixaban in patients with atrial fibrillation. N Engl J Med. 2011 Mar 3;364(9):806-17. doi: 10.1056/NEJMoa1007432. Epub 2011 Feb 10. PMID 21309657
- [Background] Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, Al-Khalidi HR, Ansell J, Atar D, Avezum A, Bahit MC, Diaz R, Easton JD, Ezekowitz JA, Flaker G, Garcia D, Geraldes M, Gersh BJ, Golitsyn S, Goto S, Hermosillo AG, Hohnloser SH, Horowitz J, Mohan P, Jansky P, Lewis BS, Lopez-Sendon JL, Pais P, Parkhomenko A, Verheugt FW, Zhu J, Wallentin L; ARISTOTLE Committees and Investigators. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011 Sep 15;365(11):981-92. doi: 10.1056/NEJMoa1107039. Epub 2011 Aug 27. PMID 21870978
- [Background] Herzog CA, Asinger RW, Berger AK, Charytan DM, Diez J, Hart RG, Eckardt KU, Kasiske BL, McCullough PA, Passman RS, DeLoach SS, Pun PH, Ritz E. Cardiovascular disease in chronic kidney disease. A clinical update from Kidney Disease: Improving Global Outcomes (KDIGO). Kidney Int. 2011 Sep;80(6):572-86. doi: 10.1038/ki.2011.223. Epub 2011 Jul 13. PMID 21750584
- [Derived] Pokorney SD, Chertow GM, Al-Khalidi HR, Gallup D, Dignacco P, Mussina K, Bansal N, Gadegbeku CA, Garcia DA, Garonzik S, Lopes RD, Mahaffey KW, Matsuda K, Middleton JP, Rymer JA, Sands GH, Thadhani R, Thomas KL, Washam JB, Winkelmayer WC, Granger CB; RENAL-AF Investigators. Apixaban for Patients With Atrial Fibrillation on Hemodialysis: A Multicenter Randomized Controlled Trial. Circulation. 2022 Dec 6;146(23):1735-1745. doi: 10.1161/CIRCULATIONAHA.121.054990. Epub 2022 Nov 6. PMID 36335914

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who met protocol inclusion criteria were enrolled (randomized 1:1 apixaban and warfarin) at clinical sites across the United States.
Groups:
- Apixaban: apixaban 5 mg twice daily (apixaban 2.5 mg twice daily for selected patients; >= 80 years old or dry body weight/hemodialysis target body weight <= 60 kg)
  apixaban: oral anticoagulant
- Warfarin: warfarin as prescribed by participant's provider dose adjusted to target International Normalized Ratio (INR) of 2-3
  warfarin: oral anticoagulant
Period: Overall Study
Arm/Group | Apixaban | Warfarin
Started | 82 | 72
Completed | 56 | 48
Not Completed | 26 | 24
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 7 | 9
Not completed — Death | 16 | 13

BASELINE CHARACTERISTICS:
Groups:
- Warfarin: warfarin daily dose adjusted to target International Normalized Ratio (INR) of 2-3
  warfarin: oral anticoagulant
- Total: Total of all reporting groups
Arm/Group | Apixaban | Warfarin | Total
Number analyzed (Participants) | 82 | 72 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 25 | 57
  >=65 years | 50 | 47 | 97
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 22 | 56
  Male | 48 | 50 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 77 | 67 | 144
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 33 | 68
  White | 43 | 36 | 79
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 82 | 72 | 154
Weight [Mean (Standard Deviation); unit: kilograms] — Dry weight of each participant is measured in kilograms.
  kilograms | 87.6 (24.1) | 93.7 (24.9) | 90.5 (24.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing ISTH (International Society on Thrombosis and Haemostasis) Major or Clinically Relevant Non-major Bleeding
Description: Assess the safety of apixaban versus warfarin regarding ISTH major bleeding or clinically relevant non-major bleeding events in patients with NVAF (nonvalvular atrial fibrillation) and ESRD (end-stage renal disease) on hemodialysis.
  Major bleeding event is defined as:Acute clinically overt bleeding (including access site related bleeding) accompanied by 1 or more of the following: Decrease in Hgb of 2g/dL or more with overt bleeding; Transfusion of 2 or more units of packed RBCs in the setting of an overt bleeding event; Bleeding within a critical site. Hemorrhagic stroke (primary or infarction with hemorrhagic conversion) were classified as major bleeds.
  Non-major bleeding event is defined as: Acute or sub-acute clinically overt bleeding (including access site related bleeding) that does not meet criteria for major bleeding & results in Hospital admission for bleeding, physician guided medical or surgical treatment for bleeding, or change in antithrombotic therapy
Time Frame: Randomization up to Month 15/Final Visit
Population: Intent to Treat Population(ITT): Consists of all unique randomized participants regardless of their compliance with the study protocol. Participants are analyzed in the treatment group to which they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 82 | 72
Participants | 21 | 16
Statistical Analysis 1: Comparison: Apixaban vs Warfarin; Exploratory analysis due to failure to reach initial sample size: Non-inferiority (NI) null hypothesis: HR >= 1.4 (Non-inferiority); Test type: Non-Inferiority — Due to a lower recruitment rate than anticipated in the early stage of the trial, the sample size was curtailed from 760 to 230 patients. Thus, under the initial protocol assumptions, the study is considered under-powered for the two-sided upper 95% CI on the HR to rule-out the non-inferiority margin of 1.40; p = 0.321, Regression, Cox; Cox model was adjusted for prior warfarin status (naive vs experienced) and treatment (apixaban vs warfarin); Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.63 to 2.3] — Time from randomization to first occurrence of outcome was modeled. If no event, censored at earliest of: most recent date of evaluation of outcome, month 15 target (460 days + randomization date), or end of study date (July 27, 2019)
Statistical Analysis 2: Comparison: Apixaban vs Warfarin; Test type: Superiority — Exploratory analysis due to lack of achieving initial sample size; p = 0.583, Regression, Cox — If upper limit of 95% confidence interval < 1 this would be considered evidence of superiority; Cox model was adjusted for prior warfarin status (naive vs experienced) and treatment (apixaban vs warfarin); Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.63 to 2.3] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants Experiencing Stroke or Systemic Embolism
Description: Number of participants experiencing adjudicated stroke or systemic embolism.
Time Frame: Randomization up to Month 15/Final Visit
Population: Intent to Treat Population (ITT): Consists of all unique randomized participants regardless of their compliance with the study protocol. Participants are analyzed in the treatment group to which they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 82 | 72
Participants | 2 | 2

3. Secondary Outcome: Number of Participants Experiencing Mortality
Description: Evaluate mortality rates for those participants randomized to warfarin and apixaban in patients with NVAF and ESRD on hemodialysis
Time Frame: Randomization up to Month 15/Final Visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 82 | 72
Participants | 21 | 13
Statistical Analysis 1: Comparison: Apixaban vs Warfarin; Hazard ratios (apixaban vs warfarin) and 95% confidence intervals obtained using Cox model adjusted for prior warfarin status (naive vs experienced) and treatment. Time from randomization to first occurrence of the composite outcome/censoring date modeled. Those that did not experience the outcome are censored at the earliest of the following: 1) most recent date of evaluation of all of the components, 2) month 15 target (460 days + randomization date), and end of study date (July 27, 2019); Test type: Superiority; No p-value provided as analysis is considered exploratory due to study being under powered; Hazard Ratio (HR) = 1.47, 95% CI 2-sided [0.74 to 2.93]

4. Secondary Outcome: Persistence of Therapy
Description: Evaluate days between time from initiation to discontinuation of randomized therapy.
Time Frame: Randomization up to Month 15/Final Visit
Population: Consists of all unique participants who took at least one dose of the randomized study drug. Participants were analyzed as randomized.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 77 | 68
Days | 304.4 (140.0) | 279.6 (138.2)

5. Secondary Outcome: Apixaban Plasma Concentration, Cmax
Description: Evaluate the pharmacokinetics of apixaban in ESRD NVAF patients on hemodialysis. The measurement was done from 0-12 hours after the dose was given on Day 1.
Time Frame: 0-12 hours post-dose
Population: Participants in the Apixaban group who had a plasma sample collected. This outcome measure is not relevant to the Warfarin group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Apixaban 2.5 mg: Plasma apixaban concentration, Cmax for apixaban 2.5 mg
- Apixaban 5 mg: Plasma apixaban concentration, Cmax for apixaban 5mg
Arm/Group | Apixaban 2.5 mg | Apixaban 5 mg
Number analyzed (Participants) | 20 | 41
ng/mL | 59.7 (34.3) | 97.9 (37.9)

6. Secondary Outcome: Apixaban Plasma Concentration, Cmin
Description: as for outcome 5
Time Frame: 0-12 hours post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Apixaban 2.5 mg: Plasma apixaban concentration, Cmin from apixaban 2.5 mg
- Apixaban 5mg: Plasma apixaban concentration, Cmin from apixaban 5 mg
Arm/Group | Apixaban 2.5 mg | Apixaban 5mg
Number analyzed (Participants) | 20 | 41
ng/mL | 28.2 (62.1) | 49.7 (57.1)

7. Secondary Outcome: Area Under the Plasma Apixaban Concentration Curve From 0 to 12 Hours After Dose (AUCO-12)
Description: Evaluate the pharmacokinetics of apixaban in ESRD NVAF patients on hemodialysis. The measurement was done from 0 to 12 hours after dose was given on Day 1.
Time Frame: 0-12 hours post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Apixaban 2.5 mg: Plasma apixaban concentration curve from 0 to 12 hours after dose for apixaban 2.5 mg
- Apixaban 5mg: Plasma apixaban concentration curve from 0 to 12 hours after dose for apixaban 5 mg
Arm/Group | Apixaban 2.5 mg | Apixaban 5mg
Number analyzed (Participants) | 20 | 41
ng*h/mL | 507 (40.4) | 868 (44)

8. Secondary Outcome: Apixaban Pharmacodynamics, Chromogenic Factor Xa Assay
Description: Evaluate the pharmacodynamics of apixaban in ESRD NVAF patients on hemodialysis
Time Frame: Baseline: Day 3, 4, or 5; Day 28
Population: Data not collected.
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Adherence to Treatment With Apixaban or With Warfarin
Description: Measured by self-reported days of medication compliance over the last 30 days.
Time Frame: Month 15/Final Visit
Population: Participants who reported medication compliance at month 15.
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 28 | 18
Participants
  5 days or fewer | 1 | 1
  6 to 23 days | 4 | 2
  24 days or more | 23 | 15

10. Other Pre Specified Outcome: Number of Participants Experiencing Systemic Embolism
Description: Adjudicated diagnosis of systemic arterial embolism (Non-pulmonary, non-cranial events) will require a positive clinical history consistent with an acute loss of blood flow to a peripheral artery (or arteries), which is supported by evidence of embolism/thrombosis from surgical specimens, autopsy, angiography, vascular imaging, or other objective testing.
  Clinical presentation would include:
  1. Abrupt development of pain, absent pulses, pallor, and/or paresis in an extremity (at least an entire digit) without previous severe claudication or findings of severe peripheral vascular disease.
  2. Renal embolism will be diagnosed when sudden flank pain or a change in renal laboratory findings occurred.
  3. Abdominal vascular/visceral embolism was considered definite if acute abdominal symptoms or referred symptoms developed along with a change in abdominal examination or appropriate laboratory values.
Time Frame: Randomization up to Month 15/Final Visit
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 82 | 72
Participants | 0 | 0

11. Other Pre Specified Outcome: Number of Participants Experiencing Stroke
Description: Adjudcated stroke defined as a new, non-traumatic episode of focal or global neurological dysfunction of sudden onset caused by central nervous system (CNS) vascular injury as a result of hemorrhage or infarction and not due to a readily identifiable non-vascular cause (i.e. brain tumor). CNS includes brain, spinal cord and retina. The required duration of the deficit is ≥ 24 hours.
  * Events with neurologic deficit lasting for < 24 hours and an imaging modality showing evidence of an acute stroke will be counted as stroke as well.
  * A retinal ischemic event (embolism, infarction) will be considered a stroke
Time Frame: Randomization up to Month 15/Final Visit
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 82 | 72
Participants | 2 | 2

12. Other Pre Specified Outcome: Number of Participants Experiencing Stroke, Systemic Embolism, Major Bleeding or All-cause Mortality
Description: Evaluate those experiencing stroke, systemic embolism, ISTH major bleeding, or all-cause mortality for those randomized to warfarin and apixaban in patients with NVAF and ESRD on hemodialysis
  Definitions of stroke and systemic embolism are provided under the measurement description of the secondary outcomes for each individual event. Definition of major bleed is provided in outcome measurement description of the primary outcome measure.
Time Frame: Randomization up to Month 15/Final Visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 82 | 72
Participants | 27 | 29
Statistical Analysis 1: Comparison: Apixaban vs Warfarin; Hazard ratios (apixaban vs warfarin) and 95% confidence intervals obtained using Cox model adjusted for prior warfarin status (naive vs experienced) and treatment. Time from randomization to first occurrence of the composite outcome/censoring date modeled. Those that did not experience the outcome are censored at the earliest of the following: 1) most recent date of evaluation of all of the components, 2) month 15 target (460 days + randomization date), and end of stud date (July 27, 2019); Test type: Superiority; No p-value provided as analysis is considered exploratory due to study being under powered; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.67 to 2.17]

13. Other Pre Specified Outcome: Baseline Biomarkers
Description: Analysis of outcomes and treatment effect according to levels of cardiovascular biomarkers at baseline
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Informed Consent date through 30 days after permanent drug discontinuation.
Description: For the apixaban group, 79 of the 82 participants randomized were assessed for adverse events. For the warfarin group, 68 of the 72 participants randomized were assessed for adverse events. The participants that were not assessed for adverse events either died on the same day as randomization (n=1) or withdrew consent for additional follow-up on Day 1 and, therefore, were not assessed for AEs. (n=6).
Arm/Group | Apixaban | Warfarin
All-Cause Mortality (participants affected / at risk) | 21/82 | 13/72
Serious Adverse Events (participants affected / at risk) | 13/79 | 8/68
Other Adverse Events (participants affected / at risk) | 4/79 | 2/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban (N=79) | Warfarin (N=68)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular dissociation (Cardiac disorders) | 1 (1) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vena cava injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Generalized Anxiety Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterly occlusion (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban (N=79) | Warfarin (N=68)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
International normalised ratio abnormal (Investigations) | 0 (0) | 1 (5)

LIMITATIONS AND CAVEATS:
PK data are not final and are undergoing further modeling and analyses that will be reported in a separate manuscript.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT02942407/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT02942407/SAP_001.pdf